CLINICAL TRIAL: NCT00378690
Title: A Phase IIIb Randomized Study of Intermittent Versus Continuous Androgen Deprivation Therapy Using ELIGARD 22.5 mg 3-month Depot in Subjects With Relapsing and Locally Advanced Prostate Cancer Who Are Responsive to Such Therapy
Brief Title: A Phase IIIb Study of Intermittent Versus Continuous Hormone Deprivation Treatment With ELIGARD
Acronym: ICELAND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGD-EC-003; 2005-004094-25 (EudraCT Number)
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostate Specific Antigen
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Androgen Deprivation (CAD) (Active Comparator)
  Interventions: Drug: leuprorelin acetate
- Intermittent Androgen Deprivation (IAD) (Experimental)
  Interventions: Drug: leuprorelin acetate

INTERVENTIONS:
Drug: leuprorelin acetate — LHRH antagonist
  Other Names: ELIGARD 22.5 mg

SUMMARY:
Phase IIIb, Open-label, randomized, controlled multi-centre study. Induction therapy phase for 6 months where all subjects receive 2 ELIGARD depot injections. Those subjects with hormone responsive prostate cancer will be randomized and will receive either intermittent or continuous ELIGARD treatment for 36 months. Following this treatment period, subjects will enter a long-term follow-up period for 48 months.

ELIGIBILITY:
Inclusion Criteria:

At study entry (visit 1):

* Written informed consent
* Male subjects aged >=18 and <80 years old
* Locally advanced (stage T3 or T4) prostate cancer or Relapsing prostate cancer following radical prostatectomy or,Relapsing prostate cancer following radiotherapy
* Gleason score of >=6
* ECOG performance status of 0-2.
* Life expectancy at least 5 years

At randomization (visit 4):

* Two successive decreasing serum PSA levels <=1 ng/ml

Exclusion Criteria:

At study entry (visit 1):

* Any suspected second primary tumors
* Evidence of metastatic disease
* Other malignancy within the last 5 years except
* Acute spinal cord compression, uni- or bilateral ureteric obstruction
* Any concurrent biological response modifier therapy
* Concurrent chemotherapy
* Less than 1 year since any prior neoadjuvant or adjuvant hormonal therapy
* Less than 6 months since prior 5-alpha reductase inhibitor treatment
* Other concurrent hormonal therapy
* Any concurrent radiotherapy
* Testosterone at screening <= 1.7 mM or 50 ng/dL
* Clinically significant elevation of serum creatinine or liver enzymes
* Hypersensitivity to GnRH or other GnRH analogues or leuprorelin acetate
* Hypersensitivity to CASODEXâ 50 mg.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2006-03; Primary Completion 2011-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Time to PSA progression | 3 Years

SECONDARY OUTCOMES:
Overall survival | 5 Years
World Health Organization/Eastern Cooperative Oncology Group (WHO/ECOG) performance status | 3 Years
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 and QLQ-PR25 | 3 Years
Time to serum testosterone > 50 ng/dL | 3 Years
Change in progression biomarkers (some sites) | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Medical Affairs Europe, Astellas Pharma Europe Limited Hillswood Drive
Locations (60):
- Belgium (3):
  - Brussels
  - Leuven
  - Liège
- Czechia (4):
  - Bmo
  - Jablonec nad Nisou
  - Olomouc
  - Ústí nad Labem
- Finland (2):
  - Joensuu
  - Tampere
- France (15):
  - Avignon
  - Bordeaux
  - Brest
  - Caen
  - Cergy-Pontoise
  - Grenoble
  - Marseille
  - Nantes
  - Paris
  - Pierre-Bénite
  - Ploemeur
  - Rouen
  - Suresnes
  - Toulon
  - Toulouse
- Germany (9):
  - Bad Neuenaher
  - Bautzen
  - Dresden
  - Hagenow
  - Halle
  - Hettstedt
  - Leipzig
  - Neustadt in Sachsen
  - Trier
- Hungary (6):
  - Budapest
  - Kaposvár
  - Nyíregyháza
  - Szolnok
  - Tatabánya
  - Veszprém
- Italy (10):
  - Bergamo, Bergamo
  - Bologna, Bologna
  - Desio, Milano
  - Parma, Parma
  - Roma, Roma
  - Ancona
  - Bari
  - Chieti
  - Messina
  - Milan
- Russia (2):
  - Moscow
  - Saint Petersburg
- Slovakia (3):
  - Martin
  - Skalica
  - Trenčín
- Spain (6):
  - Alcorcón, Madrid
  - A Coruña
  - Barcelona
  - Granada
  - Madrid
  - Valencia

REFERENCES:
- [Derived] Tombal B, Cornel EB, Persad R, Stari A, Gomez Veiga F, Schulman C. Clinical Outcomes and Testosterone Levels Following Continuous Androgen Deprivation in Patients with Relapsing or Locally Advanced Prostate Cancer: A Post Hoc Analysis of the ICELAND Study. J Urol. 2017 Nov;198(5):1054-1060. doi: 10.1016/j.juro.2017.05.072. Epub 2017 May 25. PMID 28552710
- [Derived] Schulman C, Cornel E, Matveev V, Tammela TL, Schraml J, Bensadoun H, Warnack W, Persad R, Salagierski M, Gomez Veiga F, Baskin-Bey E, Lopez B, Tombal B. Intermittent Versus Continuous Androgen Deprivation Therapy in Patients with Relapsing or Locally Advanced Prostate Cancer: A Phase 3b Randomised Study (ICELAND). Eur Urol. 2016 Apr;69(4):720-727. doi: 10.1016/j.eururo.2015.10.007. Epub 2015 Oct 29. PMID 26520703